CLINICAL TRIAL: NCT03861689
Title: A Prospective Longitudinal Study on the Effect of Tight Control Management on Perianal Crohn's Disease
Brief Title: Tight Control Management in Perianal Crohn's Disease
Acronym: PLACE-PCD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Mak Wing Yan, Assistant Professor, Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PLACE-PCD_Protocol_20200909 v6
Record Dates: First submitted 2019-02-27; First posted 2019-03-04 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Inflammatory Bowel Diseases; Perianal Fistula
Keywords: Perianal Crohn's disease; MRI
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tight control arm (Active Comparator): Patients in the tight control arm will have additional FiLAC treatment within 24 months if the anatomy of the fistula is favourable. MRI pelvis will be performed at baseline and every 6 months. Biologic dosage will be adjusted according to MRI pelvis findings.
  Interventions: Diagnostic Test: MRI pelvis
- Control arm (No Intervention): Patients in the control arm will have management according to physician own decision.

INTERVENTIONS:
Diagnostic Test: MRI pelvis — MRI pelvis monitoring every 6 months; FiLAC to treat fistula tract within 24 months if the anatomy of the fistula is favourable
  Other Names: FiLAC
  Arms: Tight control arm

SUMMARY:
Perianal Crohn's disease (pCD) affects around one-third of patients with Crohn's disease (CD) during their disease course. It represents a distinct disease phenotype and causes significant morbidity, often requiring multiple surgical interventions. However, treatment of pCD is still challenging and unsatisfactory. Only approximately one-third of pCD patients responded to biologic treatment. Overall, medical therapy with anti-TNF could only achieve prolonged remission in 30-40% of pCD cases. At the same time, surgical treatment could only lead to a favourable outcome in around 50% of patients with a higher recurrence rate in patients with complex than in simple fistulae. Recently, combination of optimal medical therapy with surgical therapy (drainage of sepsis and insertion of seton), with radiological guidance, has been suggested as the standard management so as to improve the outcomes of complex pCD.

Magnetic resonance imaging (MRI) is considered to be the gold standard imaging technique for perianal CD. It can visualise the anal sphincter and the pelvic floor muscles, as well as the fistula tracts and abscesses. Previous studies using MRI to monitor treatment response to anti-TNF revealed that radiological healing lagged behind clinical remission by a median of 12 months and that long-term maintenance therapy is probably required to prevent recurrence despite a clinically healed external opening. Therefore, we hypothesize that serial monitoring with MRI is important.

Recently, there has been some advance in the surgical treatment of perianal Crohn's disease. FiLaCTM uses a radial-emitting disposable laser fibre for endofistular therapy. Recent systemic review and meta-analysis showed that the primary success rate was 73.3% (11/15) in patients with perianal Crohn's fistula.

There has been breakthrough in the management of luminal Crohn's disease. The CALM study has showed that timely escalation of anti-TNF on the basis of clinical symptoms combined with biomarkers in patients with luminal Crohn's disease resulted in better clinical and endoscopic outcomes than symptom-driven decision alone. It is unsure whether this approach is also applicable to patients with perianal Crohn's disease.

DETAILED DESCRIPTION:
Perianal Crohn's disease (pCD) affects around one-third of patients with Crohn's disease (CD) during their disease course. It represents a distinct disease phenotype and causes significant morbidity, often requiring multiple surgical interventions. The presence of pCD causes significant burden to patients. The risk of developing perianal fistulae depends on disease location and is most commonly seen in colonic disease with rectal involvement. Perianal fistulae have been reported in 12% of subjects with small intestinal CD, 15% with ileocolonic CD, 41% with colonic CD without rectal involvement and 92% of those with colonic CD with rectal involvement. Persistently high CRP level > 31 was recently found to be independently associated with subsequent development of perianal fistula in CD patients. Besides, male gender, those who have a younger age of onset of CD, non-Caucasians and Sephardic (as opposed to Ashkenazi) Jews are all at higher risk of developing pCD.

However, treatment of pCD is still challenging and unsatisfactory. Antibiotics including metronidazole and ciprofloxacin, thiopurines and other immunomodulators failed to show radiological healing of anal fistulas. Approximately one-third of pCD patients responded to biologic treatment. The ACCENT II trial is the first double blind RCT that demonstrates the benefit of infliximab maintenance in fistulising Crohn's disease. At week 54, complete absence of draining fistulae was noted in 36% of patients in the infliximab maintenance group, compared to 19% in the placebo group. (p=0.009) There are also evidence that maintenance infliximab therapy could reduce hospitalisation, surgeries and procedures in fistulising Crohn's disease. In the CHARM study, 30% of patients with fistulae treated with adalimumab had complete fistulae closure, and this increased to 33% at 56 weeks compared with 13% in the placebo group. However, the risk of recurrence is high. Only 34% of patients remained free of relapse after one year of cessation.

Up till now, there are still no clear predictors, which can predict the response to anti-TNF therapy except the presence of proctitis. Presence of proctitis has been shown to be a poor predictor of response to anti-TNF therapy. Recently, A.J. Yarur et al. reported that patients with pCD who achieved remission had higher infliximab trough level compared to those with active fistulae [15.8 vs. 4.4 lg/mL, respectively (P < 0.0001)], and those who developed anti-infliximab antibodies had a lower chance of achieving fistula healing (OR: 0.04 [95%CI: 0.005-0.3], P < 0.001). An infliximab level of ≥10.1 µg/mL is associated with fistula healing [OR: 3.9 (95%CI: 1.34-11.8) P = 0.012]. Another, retrospective study by Davidov et. al, showed that infliximab levels at week 2 and 6 were significantly associated with fistula response at week 14 and 30. Infliximab levels of 9.25µg/mL at week 2 and 7.25 µg/mL at week 6 could best predict response to treatment.

Overall, medical therapy with anti-TNF could only achieve prolonged remission in 30-40% of pCD cases. At the same time, surgical treatment could only lead to a favourable outcome in around 50% of patients with a higher recurrence rate in patients with complex than in simple fistulae. Recently, combination of optimal medical therapy with surgical therapy (drainage of sepsis and insertion of seton), with radiological guidance, has been suggested as the standard management so as to improve the outcomes of complex pCD. An earlier study in 2003 revealed that the combination of seton placement and infliximab results in an earlier initial response (100% vs. 82.6%, p=0.014), lower recurrence rates (44% vs. 79%, p=0.001) and longer time to relapse (13.5 months vs. 3.6 months, p=0.0001) than infliximab alone. Further studies in Japan and France evaluating the efficacy of combination of seton insertion and infliximab also yielded positive results with higher chance of fistulae closure. A recent systemic review and meta-analysis of 24 studies by Yassin et al. revealed that combination therapy led to higher complete remission rate compared with single therapy (52% vs. 43%).33 Overall, long-term infliximab therapy with combined medical and surgical management produced clinical remission in 36-58%.

Magnetic resonance imaging (MRI) is considered to be the gold standard imaging technique for perianal CD. It can visualise the anal sphincter and the pelvic floor muscles, as well as the fistula tracts and abscesses. Previous studies using MRI to monitor treatment response to anti-TNF revealed that radiological healing lagged behind clinical remission by a median of 12 months and that long-term maintenance therapy is probably required to prevent recurrence despite a clinically healed external opening. Therefore, investigators hypothesize that serial monitoring with MRI is important.

Recently, there has been some advance in the surgical treatment of perianal Crohn's disease. FiLaCTM uses a radial-emitting disposable laser fibre for endofistular therapy. Recent systemic review and meta-analysis showed that the primary success rate was 73.3% (11/15) in patients with perianal Crohn's fistula.

There has been breakthrough in the management of luminal Crohn's disease. The CALM study has showed that timely escalation of anti-TNF on the basis of clinical symptoms combined with biomarkers in patients with luminal Crohn's disease resulted in better clinical and endoscopic outcomes than symptom-driven decision alone. It is unsure whether this approach is also applicable to patients with perianal Crohn's disease.

Therefore, investigators hypothesize that more proactive treatment with treating to target "Radiological healing on MRI" is associated with better outcome and the combination of examination under anesthesia with drainage of perianal abscess and together with FiLaCTM of the fistula will lead to better outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Confirmed diagnosis of perianal Crohn's disease
* On biologics or will start biologics

Exclusion Criteria:

* Patients who have perianal fistula due to causes other than Crohn's disease
* Patients who have allergic reaction / contraindications to anti-TNF
* Patients who have active cancer
* Patients who have contraindications for MRI
* Known pregnancy

For patients who refuse to participate in the tight monitoring arm, they will be consented and recruited to the control arm for comparison.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-01-12 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in the disease activity in patients with perianal Crohn's disease | 24 months
  Change in the proportion of patients with perianal Crohn's disease achieving clinical remission under tight monitoring using MRI guidance compared to standard care

SECONDARY OUTCOMES:
Number of pCD patients achieving closure of external fistula opening with FiLAC | 24 months
  Number of patients achieving closure of external fistula opening after FiLaC treatment
Proportion of pCD patients requiring proctectomy, defunctioning surgery | 24 months
  Proportion of pCD patients requiring proctectomy, defunctioning surgery
Number of surgeries required for perianal Crohn's disease | 24 months
  Number of surgeries required for perianal Crohn's disease in patients undergoing tight monitoring and that in the control group
Side effects profile | 24 months
  Number of patients with treatment-related adverse events in the tight monitoring model

OTHER OUTCOMES:
Number of patients with adverse events associated with FiLAC treatment | 24 months
  Number of patients with adverse events associated with FiLAC treatment

CONTACTS AND LOCATIONS:
Overall Officials: Wing Yan Mak, MRCP, Principal Investigator — Prince of Wales Hospital
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ardizzone S, Porro GB. Perianal Crohn's disease: overview. Dig Liver Dis. 2007 Oct;39(10):957-8. doi: 10.1016/j.dld.2007.07.152. Epub 2007 Aug 27. No abstract available. PMID 17723323
- [Background] Beaugerie L, Seksik P, Nion-Larmurier I, Gendre JP, Cosnes J. Predictors of Crohn's disease. Gastroenterology. 2006 Mar;130(3):650-6. doi: 10.1053/j.gastro.2005.12.019. PMID 16530505
- [Background] Hellers G, Bergstrand O, Ewerth S, Holmstrom B. Occurrence and outcome after primary treatment of anal fistulae in Crohn's disease. Gut. 1980 Jun;21(6):525-7. doi: 10.1136/gut.21.6.525. PMID 7429313
- [Background] Wiese DM, Schwartz DA. Managing Perianal Crohn's Disease. Curr Gastroenterol Rep. 2012 Apr;14(2):153-61. doi: 10.1007/s11894-012-0243-y. PMID 22302507
- [Background] Schwartz DA, Loftus EV Jr, Tremaine WJ, Panaccione R, Harmsen WS, Zinsmeister AR, Sandborn WJ. The natural history of fistulizing Crohn's disease in Olmsted County, Minnesota. Gastroenterology. 2002 Apr;122(4):875-80. doi: 10.1053/gast.2002.32362. PMID 11910338
- [Background] Tang LY, Rawsthorne P, Bernstein CN. Are perineal and luminal fistulas associated in Crohn's disease? A population-based study. Clin Gastroenterol Hepatol. 2006 Sep;4(9):1130-4. doi: 10.1016/j.cgh.2006.06.021. Epub 2006 Aug 14. PMID 16905369
- [Background] Cosnes J, Cattan S, Blain A, Beaugerie L, Carbonnel F, Parc R, Gendre JP. Long-term evolution of disease behavior of Crohn's disease. Inflamm Bowel Dis. 2002 Jul;8(4):244-50. doi: 10.1097/00054725-200207000-00002. PMID 12131607
- [Background] Karban A, Itay M, Davidovich O, Leshinsky-Silver E, Kimmel G, Fidder H, Shamir R, Waterman M, Eliakim R, Levine A. Risk factors for perianal Crohn's disease: the role of genotype, phenotype, and ethnicity. Am J Gastroenterol. 2007 Aug;102(8):1702-8. doi: 10.1111/j.1572-0241.2007.01277.x. Epub 2007 May 17. PMID 17509030
- [Background] Thia KT, Mahadevan U, Feagan BG, Wong C, Cockeram A, Bitton A, Bernstein CN, Sandborn WJ. Ciprofloxacin or metronidazole for the treatment of perianal fistulas in patients with Crohn's disease: a randomized, double-blind, placebo-controlled pilot study. Inflamm Bowel Dis. 2009 Jan;15(1):17-24. doi: 10.1002/ibd.20608. PMID 18668682
- [Background] Pearson DC, May GR, Fick GH, Sutherland LR. Azathioprine and 6-mercaptopurine in Crohn disease. A meta-analysis. Ann Intern Med. 1995 Jul 15;123(2):132-42. doi: 10.7326/0003-4819-123-2-199507150-00009. PMID 7778826
- [Background] Prefontaine E, Macdonald JK, Sutherland LR. Azathioprine or 6-mercaptopurine for induction of remission in Crohn's disease. Cochrane Database Syst Rev. 2010 Jun 16;(6):CD000545. doi: 10.1002/14651858.CD000545.pub3. PMID 20556747
- [Background] Sands BE, Anderson FH, Bernstein CN, Chey WY, Feagan BG, Fedorak RN, Kamm MA, Korzenik JR, Lashner BA, Onken JE, Rachmilewitz D, Rutgeerts P, Wild G, Wolf DC, Marsters PA, Travers SB, Blank MA, van Deventer SJ. Infliximab maintenance therapy for fistulizing Crohn's disease. N Engl J Med. 2004 Feb 26;350(9):876-85. doi: 10.1056/NEJMoa030815. PMID 14985485
- [Background] Lichtenstein GR, Yan S, Bala M, Blank M, Sands BE. Infliximab maintenance treatment reduces hospitalizations, surgeries, and procedures in fistulizing Crohn's disease. Gastroenterology. 2005 Apr;128(4):862-9. doi: 10.1053/j.gastro.2005.01.048. PMID 15825070
- [Background] Colombel JF, Sandborn WJ, Rutgeerts P, Enns R, Hanauer SB, Panaccione R, Schreiber S, Byczkowski D, Li J, Kent JD, Pollack PF. Adalimumab for maintenance of clinical response and remission in patients with Crohn's disease: the CHARM trial. Gastroenterology. 2007 Jan;132(1):52-65. doi: 10.1053/j.gastro.2006.11.041. Epub 2006 Nov 29. PMID 17241859
- [Background] Domenech E, Hinojosa J, Nos P, Garcia-Planella E, Cabre E, Bernal I, Gassull MA. Clinical evolution of luminal and perianal Crohn's disease after inducing remission with infliximab: how long should patients be treated? Aliment Pharmacol Ther. 2005 Dec;22(11-12):1107-13. doi: 10.1111/j.1365-2036.2005.02670.x. PMID 16305724
- [Background] Singh S, Ding NS, Mathis KL, Dulai PS, Farrell AM, Pemberton JH, Hart AL, Sandborn WJ, Loftus EV Jr. Systematic review with meta-analysis: faecal diversion for management of perianal Crohn's disease. Aliment Pharmacol Ther. 2015 Oct;42(7):783-92. doi: 10.1111/apt.13356. Epub 2015 Aug 11. PMID 26264359
- [Background] Lopez J, Konijeti GG, Nguyen DD, Sauk J, Yajnik V, Ananthakrishnan AN. Natural history of Crohn's disease following total colectomy and end ileostomy. Inflamm Bowel Dis. 2014 Jul;20(7):1236-41. doi: 10.1097/MIB.0000000000000072. PMID 24859297
- [Background] Bell SJ, Williams AB, Wiesel P, Wilkinson K, Cohen RC, Kamm MA. The clinical course of fistulating Crohn's disease. Aliment Pharmacol Ther. 2003 May 1;17(9):1145-51. doi: 10.1046/j.1365-2036.2003.01561.x. PMID 12752351
- [Background] Yamamoto T, Bain IM, Allan RN, Keighley MR. Persistent perineal sinus after proctocolectomy for Crohn's disease. Dis Colon Rectum. 1999 Jan;42(1):96-101. doi: 10.1007/BF02235190. PMID 10211527
- [Background] Loffler T, Welsch T, Muhl S, Hinz U, Schmidt J, Kienle P. Long-term success rate after surgical treatment of anorectal and rectovaginal fistulas in Crohn's disease. Int J Colorectal Dis. 2009 May;24(5):521-6. doi: 10.1007/s00384-009-0638-x. Epub 2009 Jan 27. PMID 19172284
- [Background] Regueiro M, Mardini H. Treatment of perianal fistulizing Crohn's disease with infliximab alone or as an adjunct to exam under anesthesia with seton placement. Inflamm Bowel Dis. 2003 Mar;9(2):98-103. doi: 10.1097/00054725-200303000-00003. PMID 12769443
- [Background] Tanaka S, Matsuo K, Sasaki T, Nakano M, Sakai K, Beppu R, Yamashita Y, Maeda K, Aoyagi K. Clinical advantages of combined seton placement and infliximab maintenance therapy for perianal fistulizing Crohn's disease: when and how were the seton drains removed? Hepatogastroenterology. 2010 Jan-Feb;57(97):3-7. PMID 20422862
- [Background] Bouguen G, Siproudhis L, Gizard E, Wallenhorst T, Billioud V, Bretagne JF, Bigard MA, Peyrin-Biroulet L. Long-term outcome of perianal fistulizing Crohn's disease treated with infliximab. Clin Gastroenterol Hepatol. 2013 Aug;11(8):975-81.e1-4. doi: 10.1016/j.cgh.2012.12.042. Epub 2013 Jan 30. PMID 23376316
- [Background] Yassin NA, Askari A, Warusavitarne J, Faiz OD, Athanasiou T, Phillips RK, Hart AL. Systematic review: the combined surgical and medical treatment of fistulising perianal Crohn's disease. Aliment Pharmacol Ther. 2014 Oct;40(7):741-9. doi: 10.1111/apt.12906. Epub 2014 Aug 13. PMID 25115149
- [Background] Adegbola SO, Sahnan K, Pellino G, Tozer PJ, Hart A, Phillips RKS, Warusavitarne J, Faiz OD. Short-term efficacy and safety of three novel sphincter-sparing techniques for anal fistulae: a systematic review. Tech Coloproctol. 2017 Oct;21(10):775-782. doi: 10.1007/s10151-017-1699-4. Epub 2017 Oct 29. PMID 29080959
- [Background] Gecse KB, Bemelman W, Kamm MA, Stoker J, Khanna R, Ng SC, Panes J, van Assche G, Liu Z, Hart A, Levesque BG, D'Haens G; World Gastroenterology Organization, International Organisation for Inflammatory Bowel Diseases IOIBD, European Society of Coloproctology and Robarts Clinical Trials; World Gastroenterology Organization International Organisation for Inflammatory Bowel Diseases IOIBD European Society of Coloproctology and Robarts Clinical Trials. A global consensus on the classification, diagnosis and multidisciplinary treatment of perianal fistulising Crohn's disease. Gut. 2014 Sep;63(9):1381-92. doi: 10.1136/gutjnl-2013-306709. Epub 2014 Jun 20. PMID 24951257
- [Result] Ng SC, Plamondon S, Gupta A, Burling D, Swatton A, Vaizey CJ, Kamm MA. Prospective evaluation of anti-tumor necrosis factor therapy guided by magnetic resonance imaging for Crohn's perineal fistulas. Am J Gastroenterol. 2009 Dec;104(12):2973-86. doi: 10.1038/ajg.2009.509. Epub 2009 Sep 15. PMID 19755971
- [Result] Yarur AJ, Kanagala V, Stein DJ, Czul F, Quintero MA, Agrawal D, Patel A, Best K, Fox C, Idstein K, Abreu MT. Higher infliximab trough levels are associated with perianal fistula healing in patients with Crohn's disease. Aliment Pharmacol Ther. 2017 Apr;45(7):933-940. doi: 10.1111/apt.13970. Epub 2017 Feb 17. PMID 28211593
- [Result] Hlavaty T, Pierik M, Henckaerts L, Ferrante M, Joossens S, van Schuerbeek N, Noman M, Rutgeerts P, Vermeire S. Polymorphisms in apoptosis genes predict response to infliximab therapy in luminal and fistulizing Crohn's disease. Aliment Pharmacol Ther. 2005 Oct 1;22(7):613-26. doi: 10.1111/j.1365-2036.2005.02635.x. PMID 16181301
- [Result] Tozer PJ, Burling D, Gupta A, Phillips RK, Hart AL. Review article: medical, surgical and radiological management of perianal Crohn's fistulas. Aliment Pharmacol Ther. 2011 Jan;33(1):5-22. doi: 10.1111/j.1365-2036.2010.04486.x. Epub 2010 Oct 29. PMID 21083581
- [Result] Colombel JF, Panaccione R, Bossuyt P, Lukas M, Baert F, Vanasek T, Danalioglu A, Novacek G, Armuzzi A, Hebuterne X, Travis S, Danese S, Reinisch W, Sandborn WJ, Rutgeerts P, Hommes D, Schreiber S, Neimark E, Huang B, Zhou Q, Mendez P, Petersson J, Wallace K, Robinson AM, Thakkar RB, D'Haens G. Effect of tight control management on Crohn's disease (CALM): a multicentre, randomised, controlled phase 3 trial. Lancet. 2017 Dec 23;390(10114):2779-2789. doi: 10.1016/S0140-6736(17)32641-7. Epub 2017 Oct 31. PMID 29096949
- [Result] Davidov Y, Ungar B, Bar-Yoseph H, Carter D, Haj-Natour O, Yavzori M, Chowers Y, Eliakim R, Ben-Horin S, Kopylov U. Association of Induction Infliximab Levels With Clinical Response in Perianal Crohn's Disease. J Crohns Colitis. 2017 May 1;11(5):549-555. doi: 10.1093/ecco-jcc/jjw182. PMID 28453755
- [Result] Tozer P, Ng SC, Siddiqui MR, Plamondon S, Burling D, Gupta A, Swatton A, Tripoli S, Vaizey CJ, Kamm MA, Phillips R, Hart A. Long-term MRI-guided combined anti-TNF-alpha and thiopurine therapy for Crohn's perianal fistulas. Inflamm Bowel Dis. 2012 Oct;18(10):1825-34. doi: 10.1002/ibd.21940. Epub 2012 Jan 4. PMID 22223472